CLINICAL TRIAL: NCT00858676
Title: Multicenter Trial on Clinical Utility of Acarbose in Patients With Ischemic Heart Disease Accompanied by Abnormal Glucose Regulation
Brief Title: Impact of Acarbose on Abnormal Glucose Regulation in Patients With Coronary Artery Disease (AAA Trial)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aichi Gakuin University (Other)
Responsible Party: Principal Investigator, Tatsuaki Matsubara, MD, PhD, professor, Aichi Gakuin University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGU-75
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes Mellitus; Impaired Glucose Tolerance; Coronary Artery Disease
Keywords: acarbose; diabetes mellitus; impaired glucose tolerance; coronary artery disease
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Coronary Artery Disease | interventions — Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acarbose (Active Comparator)
  Interventions: Drug: acarbose

INTERVENTIONS:
Drug: acarbose — 50mg acarbose 3 times a day PO. duration: one year
  Other Names: Glucobay

SUMMARY:
The objective of this trial is to investigate the effect of early treatment of glucose toxicity with acarbose, a drug to control postprandial hyperglycemia, on the occurence of cardiovascular events and the inhibition of atherosclerosis.

DETAILED DESCRIPTION:
Acarbose suppresses the postprandial increase in plasma glucose levels by inhibiting the activities of alpha-amylase and alpha-glucosidase involved in digestion and absorption of carbohydrates in the intestine. A clinical study involving patients with type 2 diabetes demonstrated that acarbose decreased the post-load glucose level and improved glycosylated hemoglobin control. A prospective study involving patients with impaired glucose tolerance (IGT) demonstrated that acarbose inhibited progression to type 2 diabetes and significantly reduced the risk of cardiovascular diseases. It has also been reported that acarbose slows increase in the intima-media thickness and inhibits the progression of atherosclerosis. A significant proportion of patients with acute coronary syndrome and those with stable angina pectoris suffer from diabetes or IGT, and their prognosis is poor.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with coronary artery disease, with type 2 diabetes or impaired glucose tolerance

Exclusion Criteria:

* Patients scheduled to undergo revascularization at the time of enrollment
* Patients who are being treated with an oral hypoglycemic drug or an insulin preparation
* Patients with a history of laparotomy of ileus
* Pre- and postoperative patients or individuals with severe infection or serious trauma
* Patients with gastrointestinal disorders such as diarrhea and vomiting
* Patients with a history of hypersensitivity to acarbose
* Pregnant or possibly pregnant women
* Patients who are judged by the attending physician to be otherwise ineligible

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
sudden cardiac death, fatal or non-fatal myocardial infarction, coronary revascularization, admission due to heart failure, fatal or non-fatal stroke | one year

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuaki Matsubara, MD, PhD, Principal Investigator — Department of Internal Medicine, School of Dentistry, Aichi Gakuin University
Locations (1):
- Dept. of Intern. Med., School of Dentistry, Aichi Gakuin University, Nagoya, Japan